CLINICAL TRIAL: NCT00520936
Title: A Phase II Study of Pemetrexed in Children With Recurrent Malignancies
Brief Title: A Study of Pemetrexed in Children With Recurrent Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10294; H3E-MC-JMHW (Other: Eli Lilly and Company); ADVL0525 (Other: Children's Oncology Group); NCT00459147 (obsolete NCT alias); NCT00739427 (obsolete NCT alias)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Osteosarcoma; Medulloblastoma; Sarcoma, Ewing's; Neuroblastoma (Measurable Disease); Neuroblastoma (Metaiodobenzylguanidine; Positive Evaluable); Rhabdomyosarcoma; Ependymoma; Non-brainstem High-grade Glioma
MeSH Terms: conditions — Osteosarcoma; Medulloblastoma; Sarcoma, Ewing; Neuroblastoma; Rhabdomyosarcoma; Ependymoma | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed (Experimental)
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 1910 milligrams per meter squared (mg/m^2) (or 60 milligrams per kilogram [mg/kg] if patient <12 months old), intravenous (IV), for 21 days x 17 cycles
  Other Names: LY 231514; Alimta

SUMMARY:
To determine the response rate of pemetrexed given every 21 days for the treatment of children with relapsed or refractory osteosarcoma, Ewing's sarcoma/peripheral primitive neuroectodermal tumors (PNET), rhabdomyosarcoma, neuroblastoma, ependymoma, medulloblastoma/supratentorial PNET or non-brain stem high-grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have osteosarcoma, Ewing's sarcoma, medulloblastoma, neuroblastoma, rhabdomyosarcoma, ependymoma or high-grade non-brainstem glioma
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance 0,1,2
* Adequate renal, liver and bone marrow function
* Patient's current disease state must be one with no known curative therapy or therapy proven to prolong survival with an acceptable quality of life

Exclusion Criteria:

* Growth factors that support platelet or white cell number or function must not have been administered within the last 7 days prior to enrollment (14 days if Neulasta)
* Patients with central nervous system (CNS) tumors who have not been on a stable or decreasing dose of dexamethasone or other corticosteroid for 7 days prior to enrollment
* Patients with uncontrolled infection
* Patients who have received pemetrexed previously
* Patients with pleural effusions or ascites

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2007-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arcadia, California, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Osteosarcoma: Pemetrexed 1910 milligrams per meters squared (mg/m^2) (or 60 milligrams per kilogram [mg/kg] if patient <12 months old)
- Ewing's Sarcoma/Peripheral Primitive Neuroectodermal Tumors; Rhabdomyosarcoma; Neuroblastoma (Measureable Disease); Neuroblastoma (Metaiodobenzylguanidine Positive Evaluable); Ependymoma; Medulloblastoma/Supratentorial Primitive Neuroectodermal Tumor; Non-Brainstem High-Grade Glioma: Pemetrexed 1910 mg/m^2 (or 60 mg/kg if patient <12 months old)
Period: Overall Study
Arm/Group | Osteosarcoma | Ewing's Sarcoma/Peripheral Primitive Neuroectodermal Tumors | Rhabdomyosarcoma | Neuroblastoma (Measureable Disease) | Neuroblastoma (Metaiodobenzylguanidine Positive Evaluable) | Ependymoma | Medulloblastoma/Supratentorial Primitive Neuroectodermal Tumor | Non-Brainstem High-Grade Glioma
Started | 10 (75 participants entered the study and 72 were enrolled and received study drug.) | 11 | 9 | 5 | 6 | 10 | 11 | 10
Completed | 10 (Study completion defined as treated until disease progression. Completed=progressive disease.) | 7 | 7 | 5 | 5 | 10 | 7 | 9
Not Completed | 0 | 4 | 2 | 0 | 1 | 0 | 4 | 1
Not completed — Physician Decision | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Toxicity Requiring Removal from Study | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osteosarcoma | Ewing's Sarcoma/Peripheral Primitive Neuroectodermal Tumors | Rhabdomyosarcoma | Neuroblastoma (Measureable Disease) | Neuroblastoma (Metaiodobenzylguanidine Positive Evaluable) | Ependymoma | Medulloblastoma/Supratentorial Primitive Neuroectodermal Tumor | Non-Brainstem High-Grade Glioma | Total
Number analyzed (Participants) | 10 | 11 | 9 | 5 | 6 | 10 | 11 | 10 | 72
Age Continuous [Mean (Standard Deviation); unit: years] | 14.94 (4.28) | 18.24 (3.35) | 8.74 (4.96) | 6.23 (2.98) | 9.62 (5.38) | 8.42 (4.59) | 12.00 (7.13) | 12.75 (5.15) | 11.96 (5.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 6 | 1 | 1 | 3 | 4 | 5 | 32
  Male | 6 | 3 | 3 | 4 | 5 | 7 | 7 | 5 | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Black or African American | 4 | 0 | 0 | 2 | 1 | 1 | 3 | 3 | 14
  White | 4 | 8 | 7 | 2 | 4 | 9 | 8 | 6 | 48
  Other | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Unknown | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 8 | 5 | 5 | 9 | 10 | 10 | 61
  Canada | 3 | 4 | 1 | 0 | 1 | 1 | 1 | 0 | 11
Karnofsky Performance Score [Number; unit: Participants] — Classifies patients according to their functional impairment. Scores range from 0-100, the lower the score, the worse the survival for most serious illnesses.
  100 - Normal no complaints; no evidence of disease 90 - Normal activity; minor signs of disease 80 - Activity with effort; some signs of disease 70 - Unable to carry on normal activity <=60 Needs increasing assistance up to Death (0)
  Participants
    100 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 3
    90 | 3 | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 9
    80 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
    70 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
    50 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
    Missing | 6 | 4 | 9 | 5 | 5 | 9 | 8 | 8 | 54
Lansky Play Score [Number; unit: Participants] — 100=fully active, normal. 90=minor restrictions in physically strenuous activity. 80=active, but tires more quickly. 70=both greater restriction of and less time spent in play activity. 60=up and around, but minimal active play; keeps busy with quieter activities. 50=gets dressed, but lies around much of the day; no active play, able to participate in all quiet play activities. 40=mostly in bed; participates in quiet activities. 30=in bed; needs assistance even for quiet play. 20=often sleeping; play entirely limited to very passive activities. 10=No play; does not get out of bed.
  Participants
    100 | 1 | 1 | 3 | 4 | 2 | 2 | 2 | 3 | 18
    90 | 1 | 3 | 3 | 1 | 1 | 2 | 3 | 4 | 18
    80 | 2 | 0 | 2 | 0 | 2 | 3 | 2 | 0 | 11
    70 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
    60 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4
    50 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Missing | 4 | 7 | 0 | 0 | 1 | 1 | 3 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Tumor Response (Response Rate)
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response = disappearance of all target lesions. Partial Response = 30% decrease in sum of longest diameter of target lesions. Response rate (percent [%])= (number of participants with complete response (CR) or partial response (PR) in stratum/number of participants in stratum)*100.
Time Frame: baseline to measured progressive disease (up to 1 year)
Population: All treated participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Osteosarcoma | Ewing's Sarcoma/Peripheral Primitive Neuroectodermal Tumors | Rhabdomyosarcoma | Neuroblastoma (Measureable Disease) | Neuroblastoma (Metaiodobenzylguanidine Positive Evaluable) | Ependymoma | Medulloblastoma/Supratentorial Primitive Neuroectodermal Tumor | Non-Brainstem High-Grade Glioma
Number analyzed (Participants) | 10 | 11 | 9 | 5 | 6 | 10 | 11 | 10
Percentage of Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Patients With Adverse Events, Discontinuations, or Deaths Possibly Due to Study Drug
Description: AdEERS= Adverse Event Expedited Reporting System; AE = adverse event. Patients may be counted in more than 1 category. Includes events that were considered possibly related to study drug (PRSD) as judged by the investigator.
Time Frame: every cycle (up to 2 years and 7 months)
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Osteosarcoma | Ewing's Sarcoma/Peripheral Primitive Neuroectodermal Tumors | Rhabdomyosarcoma | Neuroblastoma (Measureable Disease) | Neuroblastoma (Metaiodobenzylguanidine Positive Evaluable) | Ependymoma | Medulloblastoma/Supratentorial Primitive Neuroectodermal Tumor | Non-Brainstem High-Grade Glioma
Number analyzed (Participants) | 10 | 11 | 9 | 5 | 6 | 10 | 11 | 10
Participants
  >=1 AdEERs possibly related to study drug | 3 | 2 | 0 | 2 | 3 | 2 | 2 | 2
  Discontinued due to AE possibly related to drug | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
  Died on therapy possibly related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Died within 31 days of last dose of drug PRSD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacogenomics - Measure the Response of Genes Related to Toxicity
Description: The pharmacogenomics outcomes examining the correlation between the presence of the methylene tetrahydrofolate reductase gene and the presence of a polymorphism in the thymidylate synthase (TS) gene and/or gene promoter and toxicity were optional and will not be reported here. Results of this optional research may be reported in the future by the Children's Oncology Group in the peer-reviewed literature.
Time Frame: baseline
Population: The pharmacogenomics outcomes examining the correlation between the presence of the methylene tetrahydrofolate reductase gene and the presence of a polymorphism in the thymidylate synthase (TS) gene and/or gene promoter and toxicity were optional and will not be reported here.
Measure: Number; unit: Correlation coefficient
Arm/Group | Osteosarcoma | Ewing's Sarcoma/Peripheral Primitive Neuroectodermal Tumors | Rhabdomyosarcoma | Neuroblastoma (Measureable Disease) | Neuroblastoma (Metaiodobenzylguanidine Positive Evaluable) | Ependymoma | Medulloblastoma/Supratentorial Primitive Neuroectodermal Tumor | Non-Brainstem High-Grade Glioma
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Pemetrexed: Pemetrexed 1910 mg/m2 (or 60 mg/kg if patient <12 months old)
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 21/72
Other Adverse Events (participants affected / at risk) | 10/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=72)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Infection (Blood and lymphatic system disorders) | 2 (2)
Infection with normal ANC or Grade 1 (Blood and lymphatic system disorders) | 4 (4)
Leukocytes (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain: Tumor pain (Gastrointestinal disorders) | 1 (1)
Ulceration (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Flushing (General disorders) | 1 (1)
Pain: Extremity-limb (General disorders) | 1 (1)
Dyspnea (Infections and infestations) | 2 (2)
Rash/desquamation (Infections and infestations) | 1 (1)
GGT (Investigations) | 1 (1)
Albumin, serum-low (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Phosphate, serum-low (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum-low (Metabolism and nutrition disorders) | 2 (2)
Hemorrhage, CNS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypotension (Nervous system disorders) | 1 (1)
Mood alteration: Depression (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Death not associated with CTCAE term (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=72)
Infection with normal ANC or Grade 1 (Blood and lymphatic system disorders) | 2 (2)
Dermatology/Skin - Other (Cardiac disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Cardiac disorders) | 1 (1)
Thrombosis/thrombus/embolism (Cardiac disorders) | 1 (1)
Sodium, serum-low (Congenital, familial and genetic disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI: Rectum (Gastrointestinal disorders) | 1 (1)
Pain: Tumor pain (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Seizure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days